CLINICAL TRIAL: NCT02952716
Title: Treatment of Human Cord Blood Mononuclear Cell for Delayed Encephalopathy After Carbon Monoxide Poisoning
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liaocheng People's Hospital (Other)
Responsible Party: Principal Investigator, Chen shuangfeng, Central Laboratory Director, Liaocheng People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: cell therapy for neurology
Record Dates: First submitted 2016-10-02; First posted 2016-11-02 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Delayed Encephalopathy After Carbon Monoxide Poisoning
Keywords: carbon monoxide poisoning; delayed encephalopathy
MeSH Terms: conditions — Carbon Monoxide Poisoning | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Experimental): Human Cord Blood Mononuclear Cell will be slowly infusion three times,at one days, 30 days,at 60days.
  Interventions: Biological: Human cord blood mononuclear cell; Other: hyperbaric oxygen
- control group (Placebo Comparator): hyperbaric oxygen
  Interventions: Other: hyperbaric oxygen

INTERVENTIONS:
Biological: Human cord blood mononuclear cell — The patients were treated by human cord blood mononuclear cell through subarachnoid space
  Arms: intervention group
Other: hyperbaric oxygen — The patients were treated by hyperbaric oxygen

SUMMARY:
The effects and safety of Human cord blood mononuclear cell for delayed encephalopathy after carbon monoxide poisoning

DETAILED DESCRIPTION:
To evaluate the effect and mechanism of human cord blood mononuclear cell transplantation for delayed encephalopathy after carbon monoxide poisoning

ELIGIBILITY:
Inclusion Criteria:

* 35-60 years old.
* No serious infection, chronic diseases, diabetes and tuberculosis.
* Written informed consents were obtained from all subjects.
* Symptomatic Delayed Encephalopathy After Carbon Monoxide Poisoning.

Exclusion Criteria:

* The heart, liver, kidney and other viscera serious organic disease.
* Allergic constitution, clotting disorders, autoimmune diseases and tumors.
* Pregnancy.
* Moribund patient.
* History of prior brain injury.
* History of central nervous system disease.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Mini-Mental State Examination (MMSE) | Baseline, 4, 8, 12 and 24 weeks

SECONDARY OUTCOMES:
Chang from baseline in head CT | Baseline, 6 and 12 months
Cerebrospinal levels of IL-2,IL-4,IL-6,IL-10,TNF,IFN-γ，IL-17A，IL-8，IL-12p70，MIG，MCP-1(ng/ul) | Baseline, 1 and 2 months
Serum levels of IL-2,IL-4,IL-6,IL-10,TNF,IFN-γ，IL-17A，IL-8，IL-12p70，MIG，MCP-1(ng/ul) | Baseline,1 and 2 months
Change From Baseline in Activities of Daily Living (ADL) | Baseline, 4, 8, 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shuangfeng Chen, Ph.D., Study Director — Liaocheng People's Hospital
Locations (1):
- Liaocheng city people's hospital, Liaocheng, Shandong, China

IPD SHARING:
Plan to Share IPD: No